CLINICAL TRIAL: NCT03998618
Title: Telephone Support for Metastatic Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eskenazi Health (Other); Community Health Network (Other); Indiana University Health (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Catherine Mosher, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1812850942; R01CA230542 (NIH)
Record Dates: First submitted 2019-06-10; First posted 2019-06-26 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer
Keywords: psychotherapy; fatigue; quality of life
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Acceptance and Commitment Therapy; Educational Status; Palliative Care

STUDY DESIGN:
Intervention Model Description: Metastatic breast cancer patients (N = 250) will be randomly assigned in equal numbers to Acceptance and Commitment Therapy (ACT) or education/support using a stratified block randomization scheme to balance the groups by age (<65 yrs. vs. 65+ yrs.) and performance status (patient-reported Eastern Cooperative Oncology Group [ECOG] scores 0 or 1 vs. 2).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Patients in the ACT arm will learn new and more adaptive ways to respond to fatigue.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Education/Support (Active Comparator): Patients in the education/support arm will discuss their cancer-related concerns and receive education on services available in their medical center and community.
  Interventions: Behavioral: Education/Support

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Across six weekly 50-minute sessions, patients in the Acceptance and Commitment Therapy condition will practice various mindfulness exercises, clarify their values, and set specific goals consistent with their values. Sessions will incorporate discussion of patients' cancer experiences. Through in-session and home practice of skills, participants will learn new and more adaptive ways to respond to fatigue. Participants will receive handouts on session topics and a compact disc (CD) that we developed to guide mindfulness practices.
  Arms: Acceptance and Commitment Therapy
Behavioral: Education/Support — Across six weekly 50-minute sessions, patients in the education/support condition will discuss their concerns, including symptoms and other cancer-related stressors, with a therapist providing psychological support. The therapist will direct patients to resources for practical and health information and contact information for psychosocial services. Sessions will include an orientation to the patient's medical center, education regarding common cancer-related symptoms and quality-of-life concerns, and an overview of resources for addressing these concerns. The therapist will also describe resources for addressing financial concerns and methods of evaluating health information available via the Internet and other modalities. Participants will receive handouts on session topics and will be asked to review them as homework.
  Arms: Education/Support

SUMMARY:
This trial tests telephone-based Acceptance and Commitment Therapy (ACT), a type of psychotherapy, to reduce fatigue interference with activities, mood, and cognition in metastatic breast cancer (MBC) cancer patients. ACT includes mindfulness exercises (e.g., meditations, performing activities with greater awareness), identifying personal values (e.g., family, work), and engaging in activities consistent with these values. A total of 250 patients will be randomly assigned in equal numbers to either the ACT intervention or an education/support condition. Patients in both conditions will participate in six weekly 50-minute telephone sessions. Outcomes will be assessed at baseline, 2 weeks post-intervention, and 3 and 6 months post-intervention. The investigators hypothesize that ACT will lead to improved primary and secondary outcomes as compared to education/support. A demonstration of ACT's efficacy will lead to dissemination of the intervention and ultimately fulfill an unmet need in the comprehensive care of MBC patients.

DETAILED DESCRIPTION:
This trial tests the effect of telephone-based Acceptance and Commitment Therapy (ACT) on fatigue interference in metastatic breast cancer (MBC) patients (Aim 1) as well as secondary outcomes (Aim 2). This trial also examines increases in psychological flexibility as a hypothesized mediator of ACT's effect on fatigue interference (Aim 3). Finally, two core aspects of psychological flexibility (i.e., mindfulness/acceptance and commitment/behavior change processes) are examined as exploratory mediators of ACT's effect on fatigue interference. The study team will recruit MBC patients receiving care through Eskenazi Health or Indiana University (IU) Health. Potentially eligible patients will be mailed an introductory letter signed by their oncologist and the PI along with a consent form. The letter will have a number to call if they do not wish to be contacted further. A research assistant (RA) will call all prospective participants who do not opt out approximately 1 to 2 weeks after the letter is mailed. The RA will describe the study as outlined in the consent form and answer any questions. Then the RA will administer an eligibility screening to those who consent to participate. Eligible and consenting patients will complete a 35-minute baseline phone assessment. Following baseline assessments, MBC patients (N = 250) will be randomly assigned in equal numbers to ACT or education/support using a stratified block randomization scheme to balance the groups by age (<65 yrs. vs. 65+ yrs.) and performance status (patient-reported Eastern Cooperative Oncology Group [ECOG] scores 0 or 1 vs. 2). Patients in both study conditions will complete six weekly 50-minute telephone sessions with the first session occurring one week after baseline. For ACT participants, adherence to home practice during the past week will be assessed and recorded during each session. Blind interviewers will assess outcomes and potential mediators during 30-minute follow-up phone assessments at 2 weeks, 3 months, and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 3 weeks post-diagnosis of stage IV breast cancer and is receiving care at the Indiana University (IU) Simon Cancer Center, Eskenazi Health, IU Health North, IU Health Bloomington, IU Health Ball Memorial, IU Health Portland, IU Health Morgan, IU Health New Castle, IU Health Central-Fishers, another IU Health hospital or clinic, Community Health Network, or the Robert H. Lurie Comprehensive Cancer Center of Northwestern University.
* Patient is at least 18 years of age.
* Patient has adequate English fluency for completion of data collection.
* Patient has moderate to severe fatigue interference with functioning

Exclusion Criteria:

* Patient shows significant psychiatric or cognitive impairment that would preclude providing informed consent and study participation.
* Patient reports being able to do little activity on a functional status measure.
* Patient is receiving hospice care at screening.
* Patient does not have working phone service.
* Patient has hearing impairment that precludes participation.
* Male sex

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Mosher, Ph.D., Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Indiana University Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Community Health Network, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Results of this trial will be presented at professional meetings and published in peer-reviewed journals. The data set will be made available to qualified investigators within 6 months of the publication of the primary outcome paper. The data set will contain necessary identifiers, excluding those prohibited by HIPAA. The investigators will be required to sign a data use agreement and obtain Institutional Review Board (IRB) approval before receiving the data set.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data set will be made available to qualified investigators within 6 months of the publication of the primary outcome paper. Data will be available for at least 6 years.
Access Criteria: The data set and supporting information will be made available to qualified investigators to allow replication of analyses or secondary data analyses. The PI will review requests for data access. The investigators will be required to sign a data use agreement and obtain IRB approval before receiving the data set. The mechanism for data sharing will be reviewed by the IRB.

REFERENCES:
- [Derived] Mosher CE, Lee S, Addington EL, Park S, Lewson AB, Snyder S, Hirsh AT, Bricker JB, Miller KD, Ballinger TJ, Schneider BP, Storniolo AM, Newton EV, Champion VL, Johns SA. Randomized Controlled Trial of Acceptance and Commitment Therapy for Fatigue Interference With Functioning in Metastatic Breast Cancer. J Clin Oncol. 2025 Feb 20;43(6):662-671. doi: 10.1200/JCO.24.00965. Epub 2024 Oct 25. PMID 39454125

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 patients were excluded from the study before assignment to groups. Here is a list of the reasons:
  Not feeling well/health problems (2), Did not have time (5), Participation was too much work (4), Not interested in the study (1), Not eligible (1), Other (1)
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Started | 116 | 120
Completed | 97 | 91
Not Completed | 19 | 29
Not completed — Death | 7 | 11
Not completed — hospice enrollment | 3 | 3
Not completed — Not feeling well/health problems | 3 | 5
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy | Education/Support | Total
Number analyzed (Participants) | 116 | 120 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (11.4) | 59.6 (11.7) | 58.97 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 120 | 236
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 115 | 118 | 233
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 16 | 24
  White | 107 | 103 | 210
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 116 | 120 | 236
Household income [Count of Participants; unit: Participants] — Income data were collected in categories.
  Participants
    $0 to $50,999 | 45 | 46 | 91
    $51,000 to $99,999 | 29 | 35 | 64
    $100,000 or more | 33 | 33 | 66
    Missing data | 9 | 6 | 15
Years of education [Mean (Standard Deviation); unit: years] — Years of education
  years | 15.3 (2.38) | 15.2 (2.73) | 15.27 (2.56)
Time since stage IV breast cancer diagnosis [Mean (Standard Deviation); unit: years] — Collected from patient medical records at baseline
  years | 2.75 (3.62) | 2.94 (3.72) | 2.85 (3.67)
Chemotherapy [Count of Participants; unit: Participants] — Collected from patient medical records at baseline
  Participants
    Yes-chemotherapy received for breast cancer | 85 | 100 | 185
    No-chemotherapy not received for breast cancer | 31 | 20 | 51
Radiation [Count of Participants; unit: Participants] — Collected from patient medical records at baseline
  Participants
    Yes-radiation received for breast cancer | 93 | 90 | 183
    No-radiation not received for breast cancer | 23 | 30 | 53
Hormonal Therapy [Count of Participants; unit: Participants] — Collected from patient medical records at baseline
  Participants
    Yes-hormonal therapy received for breast cancer | 90 | 98 | 188
    No-hormonal therapy not received for breast cancer | 26 | 22 | 48
Targeted Therapy [Count of Participants; unit: Participants] — Collected from patient medical records at baseline
  Participants
    Yes-targeted therapy received for breast cancer | 37 | 36 | 73
    No-targeted therapy not received for breast cancer | 79 | 84 | 163

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Interference Subscale of Fatigue Symptom Inventory
Description: Seven items are rated on 11-point scales (0=no interference to 10=extreme interference) that assess the extent to which fatigue in the past week interfered with general level of activity, ability to bathe and dress, normal work activity (including housework), ability to concentrate, relations with others, enjoyment of life, and mood. The seven items are summed with higher total scores indicating greater fatigue interference. The total score range is 0 to 70. This is the primary outcome.
Time Frame: 2 weeks, 3 months, and 6 months post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 116 | 120
units on a scale
  Fatigue interference at 2 weeks post-intervention | 2.96 (1.90) | 3.66 (2.20)
  Fatigue interference at 3 months post-intervention | 3.24 (2.05) | 3.43 (2.25)
  Fatigue interference at 6 months post-intervention | 3.08 (2.32) | 3.64 (2.26)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = .018, Mixed Models Analysis — P-value for study group x time interaction. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 234. multiply imputed data were used in analyses; partial correlation = 0.12, 95% CI 2-sided [-0.01 to 0.25]

2. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Sleep-related Impairment
Description: This 8-item measure assesses the perceived interference of sleep problems with activities, mood, and cognition (e.g., difficulty concentrating or completing tasks). Each item is rated on a scale from 1 (not at all) to 5 (very much). Item #2 is reverse-scored and then the 8 items are summed with higher total scores indicating greater sleep-related impairment. The total scores are converted to T-scores with a range from 30.0 to 80.1. Higher T-scores indicate a worse outcome. The population mean for T-scores is 50 with a standard deviation of 10. This is a secondary outcome.
Time Frame: 2 weeks, 3 months, and 6 months post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 116 | 120
T-score
  Sleep-related impairment at 2 weeks post-intervention | 55.28 (4.22) | 56.26 (4.27)
  Sleep-related impairment at 3 months post-intervention | 54.27 (7.79) | 54.62 (8.91)
  Sleep-related impairment at 6 months post-intervention | 54.05 (7.95) | 54.78 (8.72)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = .037, Mixed Models Analysis — P-value for study group x time interaction. Probabilities for the secondary outcomes were Sidak adjusted for correlated multiple outcomes (adjusted probability for significance = 0.0085); degrees of freedom = 234. Multiply imputed data were used; partial correlation = 0.11, 95% CI 2-sided [-0.02 to 0.24]

3. Secondary Outcome: PROMIS Ability to Participate in Social Roles and Activities
Description: This 6-item measure assesses participants' ability to participate in social roles and activities. The items measure difficulty engaging in social and recreational activities as well as usual work (including housework). Each item is rated on a scale from 1 (never) to 5 (always) and is reverse coded. Then the six items are summed with higher total scores indicating greater ability to participate in social roles and activities. The total scores are converted to T-scores with a range from 26.7 to 65.0 with higher scores indicating a better outcome. The population mean for T-scores is 50 with a standard deviation of 10. This is a secondary outcome.
Time Frame: 2 weeks, 3 months, and 6 months post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 116 | 120
T-score
  Ability to participate in social roles and activities at 2 weeks post-intervention | 46.75 (6.79) | 46.66 (6.86)
  Ability to participate in social roles and activities at 3 months post-intervention | 47.49 (7.91) | 46.75 (8.56)
  Ability to participate in social roles and activities at 6 months post-intervention | 46.81 (8.17) | 46.10 (8.01)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = .355, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; degrees of freedom = 234. Multiply imputed data were used; partial correlation = 0.07, 95% CI 2-sided [-0.06 to 0.20]

4. Secondary Outcome: Functional Assessment of Cancer Therapy-General
Description: This 27-item measure evaluates physical, social/family, emotional, and functional quality of life. For each of the 4 subscale scores (i.e., Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being), the items are summed, multiplied by the number of items, and divided by the number of items answered, with higher scores indicating better quality of life. Items are rated on 0 to 4 scales. The physical well-being subscale is the sum of 7 items (all items reverse-coded) with a range of 0 to 28. The social/family well-being subscale is the sum of 7 items (none reverse-coded) with a range of 0 to 28. The emotional well-being subscale is the sum of 6 items (5 items reverse-coded) with a range of 0 to 24. The functional well-being subscale is the sum of 7 items (none reverse-coded) with a range of 0 to 28. This is a secondary outcome measure.
Time Frame: 2 weeks, 3 months, and 6 months post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 116 | 120
units on a scale
  Physical quality of life at 2 weeks post-intervention | 17.73 (5.06) | 16.99 (5.08)
  Physical quality of life at 3 months post-intervention | 17.34 (5.80) | 16.90 (6.07)
  Physical quality of life at 6 months post-intervention | 17.18 (6.05) | 16.54 (6.15)
  Social/family quality of life at 2 weeks post-intervention | 21.15 (4.71) | 20.58 (5.47)
  Social/family quality of life at 3 months post-intervention | 20.39 (5.38) | 20.71 (5.49)
  Social/family quality of life at 6 months post-intervention | 20.36 (5.05) | 20.72 (6.34)
  Emotional quality of life at 2 weeks post-intervention | 16.72 (4.20) | 16.24 (4.81)
  Emotional quality of life at 3 months post-intervention | 16.42 (4.53) | 16.16 (4.92)
  Emotional quality of life at 6 months post-intervention | 16.21 (4.84) | 16.79 (5.01)
  Functional quality of life at 2 weeks post-intervention | 17.84 (4.53) | 16.99 (5.39)
  Functional quality of life at 3 months post-intervention | 17.18 (4.90) | 16.85 (5.36)
  Functional quality of life at 6 months post-intervention | 17.47 (5.43) | 16.68 (5.28)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = .167, Mixed Models Analysis — P-value for study group x time interaction for physical quality of life. Probabilities for the secondary outcomes were Sidak adjusted for correlated multiple outcomes (adjusted probability for significance=0.0085); degrees of freedom = 234. Multiply imputed data were used; partial correlation = 0.08, 95% CI 2-sided [-0.04 to 0.21]
Statistical Analysis 2: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = .105, Mixed Models Analysis — P-value for study group x time interaction for social/family quality of life. Probabilities for the six secondary outcomes were Sidak adjusted for correlated multiple outcomes (adjusted probability for significance=0.0085); degrees of freedom = 234. Multiply imputed data were used; partial correlation = 0.09, 95% CI 2-sided [-0.03 to 0.22]
Statistical Analysis 3: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = .142, Mixed Models Analysis — P-value for study group x time interaction for emotional quality of life. Probabilities for the six secondary outcomes were Sidak adjusted for correlated multiple outcomes (adjusted probability for significance=0.0085); degrees of freedom = 234. Multiply imputed data were used; partial correlation = 0.09, 95% CI 2-sided [-0.04 to 0.22]
Statistical Analysis 4: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = .006, Mixed Models Analysis — P-value for study group x time interaction for functional quality of life. Probabilities for the six secondary outcomes were Sidak adjusted for correlated multiple outcomes (adjusted probability for significance=0.0085); degrees of freedom = 234. Multiply imputed data were used; partial correlation = 0.13, 95% CI 2-sided [0.01 to 0.26]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on each participant from the point of baseline until approximately 8 months post-baseline.
Arm/Group | Acceptance and Commitment Therapy | Education/Support
All-Cause Mortality (participants affected / at risk) | 7/116 | 11/120
Serious Adverse Events (participants affected / at risk) | 7/116 | 11/120
Other Adverse Events (participants affected / at risk) | 0/116 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acceptance and Commitment Therapy (N=116) | Education/Support (N=120)
Deaths (General disorders) | 7 (7) | 11 (11) — All patients had advanced cancer at the time of enrollment and the serious adverse events (deaths) were expected and unrelated to the study intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT03998618/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT03998618/ICF_000.pdf